CLINICAL TRIAL: NCT03226418
Title: A Phase II Study of the Impact of Clinicogenetic Risk-Stratified Management on Outcomes of Acute Myeloid Leukemia in Older Patients
Brief Title: Geriatric Assessment & Genetic Profiling to Personalize Therapy in Older Adults With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0179-17-FB; NCI-2017-01285 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA036727 (NIH)
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-05

CONDITIONS: Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Therapy-Related Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Decitabine; Injections; Idarubicin; CPX-351; Azacitidine; venetoclax; glasdegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I Intensive Induction and Consolidation Therapies (Experimental): Intensive Induction Therapy: Participants receive cytarabine intravenously (IV) on days 1-7 and idarubicin over 10-15 minutes on days 1-3 (7+3), or liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1, 3 and 5. Gemtuzumab or midostaurin is added to 7+3 as per the standard of care. Treatment continues for 1 course in the absence of unacceptable toxicity.
  Intensive Consolidation Therapy: Participants who go into remission, receive cytarabine IV over 1-3 hours twice daily (BID) on days 1, 3, and 5. Treatment repeats every 4 weeks for 2-4 courses in the absence of disease progression or unacceptable toxicity. Participants treated with liposome-encapsulated daunorubicin-cytarabine receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3. Treatment repeats every 5-8 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine; Drug: Idarubicin; Other: Laboratory Biomarker Analysis; Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II Low-intensity Induction and Consolidation Therapies (Experimental): Low-intensity: Participants receive venetoclax in combination with azacitidine or decitabine or other standard of care low-intensity therapy such as azacitidine or decitabine alone or in combination with fms-like tyrosine kinase 3 (FLT3) inhibitor such as midostaurin, low-dose cytarabine in combination with glasdegib. Venetoclax dose varies depending on drug interaction with anti-fungal agents. Given daily continuous for 3 or more months orally. Glasdegib dose is 100 mg oral daily.
  Decitabine intravenously (IV) over 1 - 3 hours daily for 5 - 10 days. Treatment repeats every 4 - 5 weeks for 3 or more courses in the absence of disease progression, unacceptable toxicity or receipt of allogeneic stem cell transplant. Azacitidine IV infusion over 10 to 40 minutes days 1 - 7. Treatment repeats every 4 - 5 weeks for 3 or more courses in the absence of disease progression, unacceptable toxicity or receipt of allogeneic stem cell transplant.
  Interventions: Drug: Decitabine; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Azacitidine; Drug: Venetoclax; Drug: glasdegib

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: Group I Intensive Induction and Consolidation Therapies
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Aza-TdC; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
  Arms: Group II Low-intensity Induction and Consolidation Therapies
Drug: Idarubicin — Given IV
  Other Names: 4-Demethoxydaunomycin; 4-demethoxydaunorubicin; 4-DMDR
  Arms: Group I Intensive Induction and Consolidation Therapies
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX-351; Cytarabine-Daunorubicin Liposome for Injection; Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos
  Arms: Group I Intensive Induction and Consolidation Therapies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Azacitidine — Given by infusion
  Other Names: VIDAZA
  Arms: Group II Low-intensity Induction and Consolidation Therapies
Drug: Venetoclax — oral tablet
  Other Names: Venclexta, Venclyxto
  Arms: Group II Low-intensity Induction and Consolidation Therapies
Drug: glasdegib — oral tablet
  Other Names: Daurismo
  Arms: Group II Low-intensity Induction and Consolidation Therapies

SUMMARY:
Acute myeloid leukemia (AML) is among the most common hematologic malignancies in adults and accounts for approximately 10,000 deaths in the United States every year. AML is commonly diagnosed in sixth or seventh decades of life. The management of AML is complex in older patients because of associated comorbidities, intolerance to high-dose chemotherapy and high-risk tumor biology. In real world practice, over one-third of patients aged 60 years and older do not receive initial chemotherapy for AML, consequently, only 10-20% of patients are alive at 3-5 years. Longer-term survival has not improved significantly in last few decades. Poor survival of older patients with AML may be improved with refined risk-stratification and therapy selection strategies, integration of principles of geriatric medicine, and use of effective but low intensity and novel therapies.

This study will examine the impact of clinicogenetic risk-stratified management on outcomes of acute myeloid leukemia in older participants (≥ 60 years) with newly diagnosed acute myeloid leukemia who receive clinicogenetic risk-stratified therapy allocation. Participants will receive standard of care intensive or low-intensity induction based on cytogenetic and geriatric assessment-based risk stratification. Participants will be evaluated for disease status, survival, quality of life and neurocognitive status for 90 days and then followed for a total of 2 years for survival data.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is among the most common hematologic malignancies in adults and accounts for approximately 10,000 deaths in the United States every year. AML is commonly diagnosed in sixth or seventh decades of life. The management of AML is complex in older patients because of associated comorbidities, intolerance to high-dose chemotherapy and high-risk tumor biology. The current approach for therapy selection is largely subjective based on chronological age, performance status and/or comorbidities, and does not clearly identify patients who should undergo or forego intensive chemotherapy. The outcomes of older patients with high-risk AML can improve with enhanced risk-stratification and therapy selection strategies, and with the use of low intensity combination chemotherapy in patients who are not fit to receive intensive chemotherapy.

Comprehensive geriatric assessment offers a thorough assessment of multiple health domains including comorbidities, polypharmacy, cognitive, nutritional, psychological, functional and social status. Such multidimensional assessment based on geriatric principles is an important tool that can improve risk-stratification and therapy selection in older patients. This approach provides a deeper understanding of the biological age and physical fitness of patients, and anticipated tolerance to chemotherapy. In older patients with AML, previous studies have demonstrated that comprehensive geriatric assessment uncovers significant functional impairments and predicts toxicities and overall survival. Hence, geriatric assessment is considered superior to therapy allocation based on assessment of age and performance status.

Up to 75 participants newly diagnosed with AML or AML equivalents, such as myeloid sarcoma, myelodysplastic syndrome in transition to AML or high-grade treatment-related myeloid neoplasm will be enrolled and assigned to one of two groups based on cytogenetic and geriatric assessment-based risk stratification. Group I will receive intensive induction and consolidation therapy. Participants will receive cytarabine and idarubicin or liposome-encapsulated daunorubicin-cytarabine to which gemtuzumab or midostaurin will be added for one course of treatment in the absence of disease progression or unacceptable toxicity. Participants who go into remission will then receive either cytarabine or liposome-encapsulated daunorubicin-cytarabine, depending on induction therapy, for up to 4 or 8 courses in the absence of disease progression or unacceptable toxicity. Group II will receive low-intensity induction and consolidation therapy. Participants will receive oral venetoclax and azacitidine, decitabine or alternate standard of care low-intensity therapies up to four courses in the absence of disease progression or unacceptable toxicity. Participants who achieve complete remission will then receive the above treatments for three or more courses in the absence of disease progression, unacceptable toxicity or receipt of allogeneic stem cell transplant. All participants are followed up for up to 2 years after completion of treatment.

Study objectives include determining the rate of complete remission and mortality at 90 days in participants who receive clinicogenetic risk-stratified therapy allocation, determining the rate of complete remission and mortality in participants who receive intensive versus low-intensity chemotherapy, determining proportion of participants with impairments detected by geriatric assessment, determining the percentage of older participants receiving allogeneic stem cell transplant during the study, and to assessing the overall survival at 1-year for the entire cohort of participants.

ELIGIBILITY:
Inclusion criteria:

* New diagnosis of de novo, secondary or treatment-related acute myeloid leukemia (AML), other AML equivalent such as myeloid sarcoma, myelodysplastic syndrome in transformation to AML, or high-grade treatment-related myeloid neoplasm
* 60 years of age or older
* Karnofsky Performance Status ≥60%
* Able and willingly give signed informed consent

Exclusion criteria:

* Acute promyelocytic leukemia (APL). Participants with brief exposure to all-trans retinoic acid (ATRA), arsenic trioxide (ATO) or similar product for suspected APL, who later turn out not to have APL, are eligible.
* Relapsed or refractory acute myeloid leukemia (AML) requiring salvage therapy
* Prior exposure to decitabine or azacitidine (exclusion criterion for use of decitabine or azacitidine)
* Participants requiring urgent initiation of chemotherapy for leukemia-related emergencies such as leukostasis or disseminated intravascular coagulopathy Participants will not be excluded solely based on current or prior use of debulking agent (e.g., hydroxyurea or cyclophosphamide). Prior or current use of leukapheresis will be allowed.
* Uncontrolled serious infection at enrollment. Infections are considered controlled if appropriate therapy has been instituted and, at enrollment, participants do not have signs of infection progression (e.g., hemodynamic instability attributable to sepsis, new symptoms, worsening physical signs or radiographic findings attributable to infection). Persistent fever without other signs or symptoms will not be interpreted as progressing infection.
* Uncontrolled clinically significant arrhythmia, myocardial ischemia or congestive heart failure within the past 2 weeks, that is considered a contraindication for initiation of chemotherapy by the treating physician
* Ejection fraction < 45% will be an exclusion criterion for intensive chemotherapy. These participants may receive low intensity therapy.
* Clinically significant kidney (e.g., glomerular filtration rate (GFR) ≤ 45ml/minute or creatinine of ≥2 mg/dl) or liver dysfunction [e.g., aspartate aminotransferase (AST)/alanine aminotransferase (ALT) and/or bilirubin ≥2 times upper limit of normal (ULN)] at enrollment that may prevent safe use of chemotherapy. These participants may be allowed to receive low-intensity chemotherapy. Participants with elevated bilirubin secondary to Gilbert syndrome will not be excluded.
* Any other condition that may not allow safe use of chemotherapy based on clinical judgment of treating oncologist

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2024-03-16 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vijaya R Bhatt, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhatt VR, Wichman CS, Koll TT, Fisher AL, Wildes TM, Haddadin M, Berger AM, Armitage JO, Holstein SA, Maness LJ, Gundabolu K. A Phase II Trial of Geriatric Assessment-Guided Selection of Treatment Intensity in Older Adults With AML. Am J Hematol. 2025 Jul;100(7):1163-1172. doi: 10.1002/ajh.27694. Epub 2025 Apr 29. PMID 40298352
- [Derived] Bhatt VR, Wichman C, Koll TT, Fisher AL, Wildes TM, Berger A, Armitage JO, Holstein SA, Maness LJ, Gundabolu K. Longitudinal changes in cognitive and physical function and health-related quality of life in older adults with acute myeloid leukemia. J Geriatr Oncol. 2024 Jan;15(1):101676. doi: 10.1016/j.jgo.2023.101676. Epub 2023 Nov 24. PMID 38000343
- [Derived] Bhatt VR, Wichman C, Al-Kadhimi ZS, Koll TT, Fisher AL, Mahato RI, Hyde RK, Berger A, Armitage JO, Holstein SA, Maness LJ, Gundabolu K. Integrating geriatric assessment and genetic profiling to personalize therapy selection in older adults with acute myeloid leukemia. J Geriatr Oncol. 2022 Jul;13(6):871-874. doi: 10.1016/j.jgo.2022.04.005. Epub 2022 Apr 18. PMID 35450817

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants ineligible
Groups:
- Group I: INTENSIVE INDUCTION THERAPY: Patients receive cytarabine intravenously (IV) on days 1-7 and idarubicin over 10-15 minutes on days 1-3 (7+3), or liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1, 3 and 5. Gemtuzumab or midostaurin are added to 7+3 as per the standard of care. Treatment continues for 1 course in the absence of unacceptable toxicity.
  INTENSIVE CONSOLIDATION THERAPY: Patients who go into remission, receive cytarabine IV over 1-3 hours twice daily (BID) on days 1, 3, and 5. Treatment repeats every 4 weeks for 2-4 courses in the absence of disease progression or unacceptable toxicity. Patients treated with liposome-encapsulated daunorubicin-cytarabine receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3. Treatment repeats every 5-8 weeks for 2 courses in the absence of disease progression, unacceptable toxicity.
  Cytarabine: Given IV
  Idarubicin: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Liposome-encapsulated Daunorubicin-Cytarabine: Given IV
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
- Group II: LOW-INTENSITY: Patients receive venetoclax in combination with azacitidine or decitabine or other standard of care low-intensity therapy such as azacitidine or decitabine alone or in combination with fms-like tyrosine kinase 3 (FLT3) inhibitor such as midostaurin, low-dose cytarabine in combination with glasdegib.
  Venetoclax dose varies depending on drug interaction with antifungal agents. Given daily continuous for >= 3 months orally. Glasdegib dose is 100 mg oral daily.
  Decitabine IV over 1-3 hours daily for 5-10 days. Treatment repeats every 4-5 weeks for >= 3 courses in the absence of disease progression, unacceptable toxicity or receipt of allogeneic stem cell transplant. Azacitidine IV infusion over 10 to 40 minutes days 1 -7. Treatment repeats every 4-5 weeks for >= 3 courses in the absence of disease progression, unacceptable toxicity or receipt of allogeneic stem cell transplant.
  Decitabine: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
  Azacitidine: Given by infusion
  Venetoclax: oral tablet
  glasdegib: oral tablet
Period: Overall Study
Arm/Group | Group I | Group II
Started | 8 | 65
Completed | 8 | 65
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group II: LOW-INTENSITY: Patients receive venetoclax in combination with azacitidine or decitabine or other standard of care low-intensity therapy such as azacitidine or decitabine alone or in combination with FLT3 inhibitor such as midostaurin, low-dose cytarabine in combination with glasdegib.
  Venetoclax dose varies depending on drug interaction with antifungal agents. Given daily continuous for >= 3 months orally. Glasdegib dose is 100 mg oral daily.
  Decitabine IV over 1-3 hours daily for 5-10 days. Treatment repeats every 4-5 weeks for >= 3 courses in the absence of disease progression, unacceptable toxicity or receipt of allogeneic stem cell transplant. Azacitidine IV infusion over 10 to 40 minutes days 1 -7. Treatment repeats every 4-5 weeks for >= 3 courses in the absence of disease progression, unacceptable toxicity or receipt of allogeneic stem cell transplant.
  Decitabine: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
  Azacitidine: Given by infusion
  Venetoclax: oral tablet
  glasdegib: oral tablet
- Total: Total of all reporting groups
Arm/Group | Group I | Group II | Total
Number analyzed (Participants) | 8 | 65 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 17 | 22
  >=65 years | 3 | 48 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 34 | 36
  Male | 6 | 31 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 7 | 61 | 68
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 7 | 60 | 67
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Symptom Burden [Median (Inter-Quartile Range); unit: units on a scale] — Each EORTC QLQ-C30 symptom sub-scale included here-Fatigue, Nausea/Vomiting, Pain, Dyspnoea, Insomnia, Appetite Loss, Constipation, Diarrhoea and Financial Difficulties-ranges from 0 (no symptom) to 100 (worst symptom). This instrument asks 28 questions about symptoms and their effects. Higher scores consistently indicate greater symptom burden. Multi-item scales are calculated by averaging their constituent items and then linearly transforming that mean to the 0-100 metric, while single-item scales are transformed directly without averaging.
  units on a scale | 0 [0 to 4.2] | 16.7 [0 to 50] | 16.7 [0 to 50]
Quality of Life as Measured by EORTC QLQ-C30 Version 3.0 at Baseline [Median (Inter-Quartile Range); unit: Units on a scale] — The baseline value shown represents the Global Health Status (GHS) scale of the EORTC QLQ-C30, version 3.0, which is scored from 0 (worst possible overall health/quality of life) to 100 (best possible); thus, higher scores denote better outcomes. The GHS score for each participant is calculated by taking the arithmetic mean of QLQ-C30 items 29 and 30 and then linearly transforming that mean to the 0 - 100 metric specified in the EORTC scoring manual.
  Units on a scale | 75 [50 to 85.4] | 50 [33.3 to 66.7] | 50 [33.3 to 75]
Baseline Functional Status [Median (Full Range); unit: score (0-100 scale)] — Karnofsky Performance Status (KPS) ranges from 0 to 100 in 10-point increments; higher scores indicate better functional ability. 'Full Range' reflects the observed minimum and maximum for each arm and for the overall cohort.
  score (0-100 scale) | 90 [80 to 100] | 80 [60 to 100] | 80 [60 to 100]
Baseline Functional Status Measure by Geriatric Assessment [Median (Full Range); unit: units on a scale] — Assessed using multiple tools from the geriatric assessment. Katz ADL ranges 0-6 (sum of six basic ADLs scored 0 = dependent, 1 = independent); higher = better basic self-care. Lawton IADL ranges 0-8 (sum of eight instrumental tasks, same 0/1 scoring); higher = better community functioning. SPPB ranges 0-12, adding three test sub-scores (balance, gait speed, chair stands each 0-4); higher = better lower-extremity performance. Each tool is interpreted on its own; no composite score is generated.
  units on a scale
    Katz ADL Index | 6 [6 to 6] | 6 [5 to 6] | 6 [5 to 6]
    Lawton IADL Index | 8 [8 to 8] | 8 [8 to 8] | 8 [8 to 8]
    SPPB | 11 [10 to 11] | 7 [3 to 9] | 7 [3 to 11]
Neurocognitive Status by MoCA at Baseline [Median (Full Range); unit: units on a scale] — The Montreal Cognitive Assessment (MoCA) is scored from 0 to 30, where higher scores reflect better cognition. Standard cut-points are ≥ 26 = normal, 18 - 25 = mild cognitive impairment, 10 - 17 = moderate impairment, and < 10 = severe impairment; no additional weighting or transformations are applied-the final score is the direct sum of item points across the 10 cognitive domains assessed.
  units on a scale | 28 [26 to 29] | 23 [21 to 24] | 23 [21 to 29]

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete Remission and Mortality in the Entire Cohort of Older Patients
Description: All analyses will be performed based on intent-to-treat principle. The method of inversion will be used to generate an interval estimate for the proportion of 90-day mortality.
Time Frame: At 90 days
Population: "It was pre-specified to report for the entire cohort as a whole in this Outcome Measure. Results for each Arm/Group are pre-specified to be reported separately in Outcome Measure 2,"
Measure: Number; unit: percentage of subjects
Groups:
- Entire Cohort: Includes entire study cohort of older adults.
Arm/Group | Entire Cohort
Number analyzed (Participants) | 73
percentage of subjects
  90-Day Mortality | 21.9
  Remission | 52.0

2. Secondary Outcome: Rate of Complete Remission and Mortality in Subsets of Older Patients Who Receive Intensive and Low-intensity Chemotherapy
Description: as for outcome 1
Time Frame: At 90 days
Reporting Status: Not Posted, anticipated posting 2025-10

3. Secondary Outcome: Baseline Functional Status Measure by Geriatric Assessment
Description: Will assess the impact of baseline functional status on the rate of complete remission and mortality.
Time Frame: At 90 days
Reporting Status: Not Posted, anticipated posting 2025-10

4. Secondary Outcome: Baseline Functional Status
Description: Will evaluate the influence of baseline functional status on the quality of life and neurocognitive status. The association between categories of functional status and quality of life will be explored using analysis of variance (ANOVA); if assumptions of ANOVA fail, Kruskal Wallis will be used. The association between functional status (fit or vulnerable) and neurocognitive status (< 25 or 26 or higher) will be explored using a chi-square test. A generalized linear mixed model will be utilized to evaluate changes in quality of life over time. The proportion (and associated 95% confidence interval) of patients with definitely or probably modifiable impairments will be presented.
Time Frame: Up to 90 days
Reporting Status: Not Posted, anticipated posting 2025-10

5. Secondary Outcome: Symptom Burden
Description: Symptom burden will be determined using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C-30 (EORTC QLQ-C30) at four time points. This instrument asks 28 questions about symptoms and their effects which are scored 1 to 4. Higher scores indicate worse symptoms and effects. Two additional questions ask about overall health and quality of life during the past week and are scored 1 to 7. Higher scores indicate better weekly health and quality of life.
Time Frame: Baseline (diagnosis), 10, 30 and 90 days following initiation of chemotherapy
Reporting Status: Not Posted, anticipated posting 2025-10

6. Secondary Outcome: Mortality at 90 Days
Description: Mortality at 90 days will be calculated from date of diagnosis to date of death due to any cause within 90 days from diagnosis.
Time Frame: Up to 90 days from diagnosis
Measure: Number; unit: participants
Arm/Group | Group I | Group II
Number analyzed (Participants) | 8 | 65
participants | 1 | 15

7. Secondary Outcome: Quality of Life as Measured by European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire
Description: The European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30), Version 3.0, will be given at several time points in follow-up after completion of treatment. The instrument assesses cancer patients' physical, psychological and social functions. The questionnaire is composed of multi-item scales and single items.
  A linear transformation is used to standardise the raw score, so that scores range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms. The scores will be utilized to determine quality of life status will be used to evaluate changes in quality of life over time.
Time Frame: Several time points after completion of treatment, up to 2 years
Reporting Status: Not Posted, anticipated posting 2025-10

8. Secondary Outcome: Neurocognitive Status as Measured by the Montreal Cognitive Assessment (MoCA)
Description: The Montreal Cognitive Assessment (MoCA) will be given at several time points in follow-up after completion of treatment. The instrument assesses different cognitive domains, including attention, visuospatial skills, executive functions, memory, language, and abstract thinking. Each task has a specific scoring guide, with points awarded based on performance. Composite scores of 26-30 generally indicates normal cognitive function, 18-25 suggests mild cognitive impairment, 10-17 indicates moderate impairment, and scores below 10 point to severe cognitive impairment.
Time Frame: Several time points after completion of treatment, up to 2 years
Reporting Status: Not Posted, anticipated posting 2025-10

ADVERSE EVENTS:
Time Frame: Ongoing from initiation of study drug until 30 days after last administration of study drug, up to 20 weeks
Arm/Group | Group I | Group II
All-Cause Mortality (participants affected / at risk) | 1/8 | 15/65
Serious Adverse Events (participants affected / at risk) | 5/8 | 41/65
Other Adverse Events (participants affected / at risk) | 7/8 | 65/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (N=8) | Group II (N=65)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 19 (20)
Fever (General disorders) | 2 (2) | 3 (5)
Gallbladder infection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter-related infection (Infections and infestations) | 0 (0) | 2 (2)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 1 (1)
Death NOS (General disorders) | 0 (0) | 4 (4)
Investigations - Other (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 2 (2)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal/Urinary disorders - Other (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 2 (3)
Nervous system disorders - Other (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (3)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (N=8) | Group II (N=65)
Anemia (Blood and lymphatic system disorders) | 7 (7) | 65 (65)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (7) | 65 (65)
Platelet count decreased (Blood and lymphatic system disorders) | 7 (7) | 65 (65)
Neutrophil count decreased (Blood and lymphatic system disorders) | 7 (7) | 63 (63)
White blood cell decreased (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Blood bilirubin increased (Investigations) | 2 (2) | 3 (5)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT03226418/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT03226418/ICF_001.pdf